CLINICAL TRIAL: NCT04429880
Title: A Study of Oxytocin Pharmacokinetics After Intravenous Administration in Healthy Subjects and Advanced Knee Arthritis Subjects
Brief Title: A Study of Oxytocin PK After IV Administration in Healthy Subjects and Advanced Knee Arthritis Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated; no subjects enrolled. A replacement study will be submitted
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00065787
Record Dates: First submitted 2020-06-04; First posted 2020-06-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Each participant will receive the same dose of oxytocin 17 micrograms via a 10 minute intravenous infusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oxytocin (Experimental): Oxytocin 17 micrograms infusion over 10 minutes
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin given by intravenous route
  Other Names: Pitocin

SUMMARY:
The main purpose of this study is to sample the blood and calculate the pharmacokinetics (PK) of oxytocin.

This is an unblinded, sequential study of subjects, all of whom will receive an intravenous (IV) infusion of oxytocin (naturally occurring hormone that is made in the brain) with blood samples taken thereafter in order to create a formula to describe the concentrations of oxytocin in the blood over time (pharmacokinetics).

In this study healthy volunteers and people with knee arthritis so severe that they may need joint replacement are recruited for a one day study. Each study participant will have 2 IV catheters placed (one in each arm). After placement of the IV catheters and infusion of oxytocin will be given over a 10 minute period. Blood samples will be taken before the infusion begins and several times during and after the infusion. The blood will be drawn through the second IV catheter.

The investigators will also do some tests to get a rough idea of how oxytocin changes perceptions on the skin and how this relates to the amount of oxytocin in the blood at the same time. Two kinds of perceptions will be studied. First, the investigators will study a painful perception by placing a probe on the skin and heating it to 113 degrees Fahrenheit for 5 minutes. Each study participant will score any pain that is experienced on a 0 to 10 scale, and most people find that pain rises during the 5 minutes, but remains mild, usually around only 1 or 2 on the 0 to 10 scale. Secondly, the investigators will study the perception of vibration, like one feels with a tuning fork on the skin. For this the investigators will put a controlled vibration device on the arm and start the vibration at such a high frequency (1000 times per second) that it cannot be felt as vibrating. The investigators will slow the frequency until the study participant first feels vibration, then turn off the machine and record this threshold frequency where it is first felt.

DETAILED DESCRIPTION:
This is an unblinded, sequential study of subjects; all participants will receive an infusion of oxytocin with blood samples taken thereafter in order to create a formula to describe the concentrations of oxytocin in the blood over time (pharmacokinetics). In this study healthy volunteers and people with knee arthritis so severe that they may need joint replacement are recruited for a one day study. Participants will come to the Clinical Research Unit (CRU) and have two IVs inserted; one in each arm. Participants will get a 10 minute infusion through one of the IVs of oxytocin and blood will be taken several times over the next 120 minutes and the amount of oxytocin measured in the blood samples. This information will be analyzed by another group at Stanford University in the Pharmacokinetics/Pharmacodynamics (PK/PD) Core part of this application. Mathematics will be utilized to fit the amount of oxytocin over time as it disappears from blood to a formula, called pharmacokinetics. The effect of subject age, sex, race, ethnicity and weight on the pharmacokinetics of oxytocin will be tested for, since these things can affect how quickly drugs circulate in the blood and are important to better adjust the dose of drug to the individual.

The main purpose of this study is to sample the blood and calculate the pharmacokinetics of oxytocin. Investigators will also do some tests to get a rough idea of how oxytocin changes perceptions on the skin and how this relates to the amount of oxytocin in the blood at the same time. Two kinds of perceptions will be studied. In the first the study team will study a painful perception by placing a probe on the skin and heating it to 113 degrees F for 5 minutes. Subjects will score any pain felt on a 0 to 10 scale, and most people find that pain rises during the 5 minutes, but remains mild, usually around only 1 or 2 on the 0 to 10 scale. In the second, the study team will study the perception of vibration, like one feels with a tuning fork on the skin. For this the study team will put a controlled vibration device on the arm and start the vibration at such a high frequency (1000 times per second) that it cannot be felt as vibrating. The study team will slow the frequency until the subject first feels vibration, then turn off the machine and record this threshold frequency where the participant first feels it. Investigators do these two tests because they test the response of two kinds of nerve fibers - pain fibers and touch fibers - which oxytocin might affect in different ways. With this information investigators will compare the amount of oxytocin in blood over time to its effects on pain and vibration over time using mathematics.

The research participants will not benefit from this study, but the knowledge investigators get will be important not only to adjust oxytocin dose to individuals, but to study its possible effects on pain in a very standardized way. The sample size chosen is needed to get an accurate estimate for the parameters in the pharmacokinetic model for the population, not just the subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
* 2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
* 3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication. For knee arthritis subjects, normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
* 4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

* 1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
* 2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
* 3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
* 4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of oxytocin in serum | 1 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 2 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 5 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 10 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 12 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 15 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 20 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 30 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 60 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 90 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.
Pharmacokinetics of oxytocin in serum | 120 minute after oxytocin infusion initiated
  Blood will be sampled at specified intervals during and after the infusion. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration.

SECONDARY OUTCOMES:
Pharmacodynamics of heat pain after oxytocin | 30 minutes after oxytocin infusion initiated
  Pain at the end of 5 minutes of heating the skin to 45 degrees Celsius will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain after oxytocin | 60 minutes after oxytocin infusion initiated
  Pain at the end of 5 minutes of heating the skin to 45 degrees Celsius will be determined,pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain after oxytocin | 90 minutes after oxytocin infusion initiated
  Pain at the end of 5 minutes of heating the skin to 45 degrees Celsius will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain after oxytocin | 120 minutes after oxytocin infusion initiated
  Pain at the end of 5 minutes of heating the skin to 45 degrees Celsius will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain after oxytocin | 180 minutes after oxytocin infusion initiated
  Pain at the end of 5 minutes of heating the skin to 45 degrees Celsius will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of vibration perception after oxytocin | 30 minutes after oxytocin infusion initiated
  Threshold frequency for detection of vibration will be determined.Verbal report on detection of vibration.
  The threshold for first feeling vibration as the frequency of the stimulus is changed will be recorded for each subject. This is done by applying the probe to the skin and reducing frequency from 1000 Hz until the subject perceives the vibration. This is repeated 3 times and the average is taken as the value
Pharmacodynamics of vibration perception after oxytocin | 60 minutes after oxytocin infusion initiated
  Threshold frequency for detection of vibration will be determined.Verbal report on detection of vibration.
  The threshold for first feeling vibration as the frequency of the stimulus is changed will be recorded for each subject. This is done by applying the probe to the skin and reducing frequency from 1000 Hz until the subject perceives the vibration. This is repeated 3 times and the average is taken as the value
Pharmacodynamics of vibration perception after oxytocin | 90 minutes after oxytocin infusion initiated
  Threshold frequency for detection of vibration will be determined.Verbal report on detection of vibration.
  The threshold for first feeling vibration as the frequency of the stimulus is changed will be recorded for each subject. This is done by applying the probe to the skin and reducing frequency from 1000 Hz until the subject perceives the vibration. This is repeated 3 times and the average is taken as the value
Pharmacodynamics of vibration perception after oxytocin | 120 minutes after oxytocin infusion initiated
  Threshold frequency for detection of vibration will be determined. Verbal report on detection of vibration.
  The threshold for first feeling vibration as the frequency of the stimulus is changed will be recorded for each subject. This is done by applying the probe to the skin and reducing frequency from 1000 Hz until the subject perceives the vibration. This is repeated 3 times and the average is taken as the value
Pharmacodynamics of vibration perception after oxytocin | 180 minutes after oxytocin infusion initiated
  Threshold frequency for detection of vibration will be determined.Verbal report on detection of vibration.
  The threshold for first feeling vibration as the frequency of the stimulus is changed will be recorded for each subject. This is done by applying the probe to the skin and reducing frequency from 1000 Hz until the subject perceives the vibration. This is repeated 3 times and the average is taken as the value

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No